CLINICAL TRIAL: NCT06315972
Title: Combining Clemastine and Aerobic Exercise to Treat Cognitive Dysfunction in Schizophrenia by Targeting Myelin Plasticity
Acronym: OligoTreat
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Lena Deller, M.Sc., LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-000054-28
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clemastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Application of double-blind add-on clemastine at a dosage of 8 mg/day (morning: 4 mg; evening: 4 mg) + aerobic exercise training 50 min 3x/week over a period of 3 months
  Interventions: Drug: clemastine (8 mg/day)
- Control intervention (Placebo Comparator): Application of double-blind add-on placebo (morning and evening) + aerobic exercise training 50 min 3x/week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: clemastine (8 mg/day) — add-on clemastine (8 mg/day) + aerobic exercise training
  Arms: Experimental intervention
Drug: Placebo — add-on placebo + aerobic exercise training
  Arms: Control intervention

SUMMARY:
Schizophrenia (SZ) is a broad clinical entity characterized by different subjective symptoms,behavioural signs, and disease course. Research has pointed to numerous biological indicators tentatively associated with neurocognitive dysfunction, brain structural and neurochemical alterations. Cognitive deficits occur as early as the prodromal phase of the illness and significantly determine its outcome. Pathophysiologically, SZ is regarded as a disconnectome disorder in which frontal and temporal brain regions are functionally disconnected, which contributes substantially to the development of cognitive dysfunction.

Impaired connectivity is related to synaptic (microconnectivity) and myelin (macroconnectivity) plasticity. With design-based stereology, a decreased number of oligodendrocytes (OLs) in the CA4 hippocampal subregion as the basis for disturbed myelination and impaired cognition, but also a decrease in the prefrontal cortex were observed. Animal studies demonstrated that clemastine enhances remyelination by increasing the differentiation of oligodendrocyte precursor cells (OPCs) and showed that aerobic exercise increases the rate of remyelination and proliferation of OPCs; this clinically meaningful effect of aerobic exercise is stronger in combination with clemastine. Furthermore, aerobic exercise improves everyday functioning, measured by the Global Assessment of Functioning (GAF) scale, and cognitive dysfunction in SZ and increases hippocampal volume, especially the volume in the hippocampal CA4 subregion. This regional volume change correlates negatively with global and cell-specific polygenic risk scores (PRSs), indicating that OPCs are involved in the genetic risk mechanisms and disturbed plasticity underlying SZ. In patients with multiple sclerosis, 90 days' administration of clemastine fumarate 10.72 mg/day, corresponding to clemastine 8 mg/day, significantly decreased the P100 latency delay of visual evoked potentials (VEPs) as a sign of myelin repair. In a bicentric, randomized, double-blind, controlled phase IIb clinical trial with a 2-arm parallel group design in patients with SZ, the study will compare the effects of aerobic exercise training plus clemastine vs. aerobic exercise training plus placebo over a period of 3 months on 1) everyday functioning and 2) working memory as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent obtained from the participant prior to performing any protocol-related procedures, including screening evaluations

  * A DSM-V diagnosis of schizophrenia or schizophrenia-spectrum disorder according to MINI interview
  * Age between 18 and 65 years EudraCT Number: 2022-000054-28 Confidential OligoTreat Study Protocol Version 2.0 06.09.2023 9 of 62
  * Total Positive and Negative Syndrome Scale (PANSS) score ≤ 75 at V0
  * Stable antipsychotic treatment dose for at least one week prior to inclusion
  * Stable CNS-active treatment substance and dose (e.g. antidepressants and mood stabilizers) for at least one week prior to inclusion
  * Female participants with reproductive potential must have a negative beta- HCG serum pregnancy test as part of the screening visit
  * Female participants with reproductive potential must have a negative serum pregnancy test within seven days prior to randomization
  * Male participants and female participants who are not capable of bearing children or who use a method of contraception that is medically approved by the health authority of the respective country at screening

Exclusion Criteria:

* Patients who are unable to give informed consent

  * Coercive treatment at the time of study inclusion
  * Treatment-naïve schizophrenia defined as cumulative treatment with an antipsychotic agent lifetime for <30 days
  * Insufficient understanding of the German language
  * Patients with primary active (moderate or severe) substance use disorder (other than nicotine) according to MINI interview (DSM-V): patients fulfilling early (>3 months) or sustained (>12 months) remission criteria and/or with low severity of substance use disorder according to MINI are eligible for the study
  * Known clinically relevant CNS disorder(s), such as epilepsy or history of seizures
  * Concomitant use of any other putative remyelinating therapy as determined by investigator
  * Co-occurrent unstable somatic condition
  * Known porphyria
  * Known narrow-angle glaucoma, stenosing peptic ulcer, pyloroduodenal obstruction, prostatic hypertrophy with urinary retention and bladder neck obstruction Current treatment with agents with strong anticholinergic properties, such as MAO-inhibitors, opioid antagonists, clozapine at the time of study inclusion
  * Known intolerance, allergy/contraindications to one of the study drugs or any of the excipients or other agents with similar chemical properties as the study drugs (such as other arylalkylamine antihistamines)
  * Clinically relevant liver and/or renal impairment (serum creatinine >1.5mg/dl or eGFR<30 ml/min/1.73 m2 at screening, AST or ALT > 2-times the upper limit of normal at screening)
  * Current treatment with macrolide-antibiotics (such as erythromycin, clarithromycine) or azole-type antimycotics
  * Clinically relevant cardiac comorbidities (i.e. Long QT-syndrome)
  * Current hypokalaemia and/or clinically relevant hyponatraemia at screening
  * Patient-reported hereditary galactose-intolerance and/or Lapp lactosedeficiency, lactose intolerance and/or glucose-galactose malabsorption
  * Pregnancy or breast-feeding
  * Concurrent enrolment in another clinical trial where the participant is receiving an IMP or participation in another clinical trial with IMP during the last 30 days before inclusion or 7 half-lives of previously used IMP, whichever is longer.
  * For the optional MRI assessments: potential MRI contraindication(s)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
change in Global Assessment of Functioning | 3 months
  change in Global Assessment of Functioning (GAF) scores from the start of the intervention period (V1.1) to primary outcome visit after 90-93 days of treatment (V2).
change in working memory performance | 3 months
  change in working memory performance assessed by the n-back test (2-back level, d-prime) from V1.1 to V2.

IPD SHARING:
Plan to Share IPD: Undecided